CLINICAL TRIAL: NCT04251559
Title: Evaluation of the Relationship Between Age at Menarche and Gestational Diabetes Mellitus
Brief Title: Evaluation of Risk Factors for Gestational Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, mehmet ozsurmeli, principal investigator, Derince Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 240785
Record Dates: First submitted 2020-01-17; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Diabetes, Gestational; Menstrual Cycle Abnormal
Keywords: menarche; gestational diabetes mellitus; cycle, menstrual
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with gestational diabetes mellitus (Active Comparator): study group
  Interventions: Other: oral glucose loading test
- healthy participants (Placebo Comparator): control group
  Interventions: Other: oral glucose loading test

INTERVENTIONS:
Other: oral glucose loading test — oral glucose loading test was performed to all participants. gestational diabetes and control group were compared in terms of menarche age.

SUMMARY:
This study examines the relationship between the age at menarche and gestational diabetes mellitus (GDM). In this retrospective study, the sample included all pregnant women diagnosed with GDM in a pregnancy polyclinic in Kocaeli, Turkey between 2014 and 2019. The sample included 373 participants: 233 in the GDM group and 140 in the control group. The groups were compared in terms of age at menarche.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with gestational diabetes

Exclusion Criteria:

* Patients with hypertension and pregestational diabetes mellitus
* Patients with rheumatologic, nephrological, and hematological diseases
* Presence of active infection,
* corticosteroid use, acetylsalicylic acid, and anticoagulant use

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 374 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Gestational diabetes mellitus risk faktors | From the 24th week of pregnancy to the delivery
  It was evaluated whether the menarche age of pregnant women with gestational diabetes was different from pregnancy without gestational diabetes.

CONTACTS AND LOCATIONS:
Overall Officials: mehmet ozsurmeli, Study Chair — Derince Training and Research Hospital
Locations (1):
- Derince Training and Research Hospital, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bellamy L, Casas JP, Hingorani AD, Williams D. Type 2 diabetes mellitus after gestational diabetes: a systematic review and meta-analysis. Lancet. 2009 May 23;373(9677):1773-9. doi: 10.1016/S0140-6736(09)60731-5. PMID 19465232
- [Background] Bratke H, Bruserud IS, Brannsether B, Assmus J, Bjerknes R, Roelants M, Juliusson PB. Timing of menarche in Norwegian girls: associations with body mass index, waist circumference and skinfold thickness. BMC Pediatr. 2017 Jun 6;17(1):138. doi: 10.1186/s12887-017-0893-x. PMID 28587648
- [Background] Chen L, Li S, He C, Zhu Y, Buck Louis GM, Yeung E, Hu FB, Zhang C. Age at Menarche and Risk of Gestational Diabetes Mellitus: A Prospective Cohort Study Among 27,482 Women. Diabetes Care. 2016 Mar;39(3):469-71. doi: 10.2337/dc15-2011. Epub 2016 Jan 26. PMID 26813668
- [Background] De Sanctis V, Rigon F, Bernasconi S, Bianchin L, Bona G, Bozzola M, Buzi F, De Sanctis C, Tonini G, Radetti G, Perissinotto E. Age at Menarche and Menstrual Abnormalities in Adolescence: Does it Matter? The Evidence from a Large Survey among Italian Secondary Schoolgirls. Indian J Pediatr. 2019 Jan;86(Suppl 1):34-41. doi: 10.1007/s12098-018-2822-x. Epub 2019 Jan 10. PMID 30628040
- [Background] DeSisto CL, Kim SY, Sharma AJ. Prevalence estimates of gestational diabetes mellitus in the United States, Pregnancy Risk Assessment Monitoring System (PRAMS), 2007-2010. Prev Chronic Dis. 2014 Jun 19;11:E104. doi: 10.5888/pcd11.130415. PMID 24945238
- [Background] Dishi M, Enquobahrie DA, Abetew DF, Qiu C, Rudra CB, Williams MA. Age at menarche, menstrual cycle characteristics and risk of gestational diabetes. Diabetes Res Clin Pract. 2011 Sep;93(3):437-42. doi: 10.1016/j.diabres.2011.07.001. Epub 2011 Aug 3. PMID 21816498
- [Background] Feng Y, Hong X, Wilker E, Li Z, Zhang W, Jin D, Liu X, Zang T, Xu X, Xu X. Effects of age at menarche, reproductive years, and menopause on metabolic risk factors for cardiovascular diseases. Atherosclerosis. 2008 Feb;196(2):590-7. doi: 10.1016/j.atherosclerosis.2007.06.016. Epub 2007 Aug 6. PMID 17675039
- [Background] Flom JD, Cohn BA, Tehranifar P, Houghton LC, Wei Y, Protacio A, Cirillo P, Michels KB, Terry MB. Earlier age at menarche in girls with rapid early life growth: cohort and within sibling analyses. Ann Epidemiol. 2017 Mar;27(3):187-193.e2. doi: 10.1016/j.annepidem.2017.01.004. Epub 2017 Jan 19. PMID 28215584
- [Background] Freedman DS, Khan LK, Serdula MK, Dietz WH, Srinivasan SR, Berenson GS; Bogalusa heart study. The relation of menarcheal age to obesity in childhood and adulthood: the Bogalusa heart study. BMC Pediatr. 2003 Apr 30;3:3. doi: 10.1186/1471-2431-3-3. Epub 2003 Apr 30. PMID 12723990
- [Background] Gilmartin AB, Ural SH, Repke JT. Gestational diabetes mellitus. Rev Obstet Gynecol. 2008 Summer;1(3):129-34. PMID 19015764
- [Background] He C, Zhang C, Hunter DJ, Hankinson SE, Buck Louis GM, Hediger ML, Hu FB. Age at menarche and risk of type 2 diabetes: results from 2 large prospective cohort studies. Am J Epidemiol. 2010 Feb 1;171(3):334-44. doi: 10.1093/aje/kwp372. Epub 2009 Dec 21. PMID 20026580
- [Background] Lakshman R, Forouhi N, Luben R, Bingham S, Khaw K, Wareham N, Ong KK. Association between age at menarche and risk of diabetes in adults: results from the EPIC-Norfolk cohort study. Diabetologia. 2008 May;51(5):781-6. doi: 10.1007/s00125-008-0948-5. Epub 2008 Mar 5. PMID 18320165
- [Background] Lakshman R, Forouhi NG, Sharp SJ, Luben R, Bingham SA, Khaw KT, Wareham NJ, Ong KK. Early age at menarche associated with cardiovascular disease and mortality. J Clin Endocrinol Metab. 2009 Dec;94(12):4953-60. doi: 10.1210/jc.2009-1789. Epub 2009 Oct 30. PMID 19880785
- [Background] Lian Q, Mao Y, Luo S, Zhang S, Tu X, Zuo X, Lou C, Zhou W. Puberty timing associated with obesity and central obesity in Chinese Han girls. BMC Pediatr. 2019 Jan 3;19(1):1. doi: 10.1186/s12887-018-1376-4. PMID 30606158
- [Background] Li H, Shen L, Song L, Liu B, Zheng X, Xu S, Wang Y. Early age at menarche and gestational diabetes mellitus risk: Results from the Healthy Baby Cohort study. Diabetes Metab. 2017 Jun;43(3):248-252. doi: 10.1016/j.diabet.2017.01.002. Epub 2017 Feb 1. PMID 28161369
- [Background] Shen Y, Hu H, D Taylor B, Kan H, Xu X. Early Menarche and Gestational Diabetes Mellitus at First Live Birth. Matern Child Health J. 2017 Mar;21(3):593-598. doi: 10.1007/s10995-016-2143-5. PMID 27456304
- [Background] Sun X, Yang L, Pan J, Yang H, Wu Y, Chen Z, Chen X, Mu L. Age at menarche and the risk of gestational diabetes mellitus: a systematic review and meta-analysis. Endocrine. 2018 Aug;61(2):204-209. doi: 10.1007/s12020-018-1581-9. Epub 2018 Mar 20. PMID 29556913
- [Background] Toulis KA, Goulis DG, Kolibianakis EM, Venetis CA, Tarlatzis BC, Papadimas I. Risk of gestational diabetes mellitus in women with polycystic ovary syndrome: a systematic review and a meta-analysis. Fertil Steril. 2009 Aug;92(2):667-77. doi: 10.1016/j.fertnstert.2008.06.045. Epub 2008 Aug 16. PMID 18710713
- [Background] Xiao Y, Chen R, Chen M, Luo A, Chen D, Liang Q, Cai Y, Chen L, Zhao X. Age at menarche and risks of gestational diabetes mellitus: a meta-analysis of prospective studies. Oncotarget. 2017 Dec 23;9(24):17133-17140. doi: 10.18632/oncotarget.23658. eCollection 2018 Mar 30. PMID 29682210